CLINICAL TRIAL: NCT05506410
Title: A Prospective Clinical Study of Hanlikang and BTK Inhibitors in the Treatment of Newly Diagnosed Mantle Cell Lymphoma
Brief Title: A Clinical Study of Hanlikang and BTK Inhibitors in the Treatment of Newly Diagnosed Mantle Cell Lymphoma
Status: Recruiting | Type: Observational
Sponsor: Zhengzhou University (Other)
Responsible Party: Principal Investigator, Mingzhi Zhang, Director of the Oncology Department, The First Affiliated Hospital of Zhengzhou University, Zhengzhou University
Other Study IDs: hnslblzlzx20220812
Record Dates: First submitted 2022-08-13; First posted 2022-08-18 (Actual); Last update posted 2022-08-18 (Actual); Status verified 2022-08

CONDITIONS: Newly Diagnosed Mantle Cell Lymphoma
MeSH Terms: interventions — Rituximab; Bendamustine Hydrochloride; Cytarabine; Prednisone

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Arms: Experimental:Rituximab、Bendamustine、Cytarabine、Prednisone （R-BAP） combined with BTK inhibitors To observe the efficacy and safety of R-BAP combined with BTK inhibitors in the treatment of newly-treated patients with mantle cell lymphoma (MCL)
  Interventions: Drug: Rituximab

INTERVENTIONS:
Drug: Rituximab — Young patients (< 65 years of age) were treated with R-BAP for 6 cycles (efficacy was assessed every 2 cycles, and adverse events were recorded), together with oral ibrutinib, followed by oral ibrutinib for 1 year after chemotherapy (efficacy was assessed every 3 months). Elderly patients (≥65 years of age) received 4 cycles of R-BAP (efficacy assessed every 2 cycles, and adverse reactions recorded), followed by 4 cycles of rituximab consolidation (efficacy assessed every 2 cycles) and 1 year of oral zanubrutinib (efficacy assessed every 3 months).
  Other Names: Bendamustine; Cytarabine; Prednisone; BTK inhibitors

SUMMARY:
An open-label, single-arm, multicenter, prospective clinical study of Hanlikang and BTK inhibitors in the treatment of newly diagnosed mantle cell lymphoma

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-70, ECOG score 0-2;
2. Estimated survival time >6 months;
3. Mantle cell lymphoma was confirmed by pathology.
4. Acceptable hematological indexes without chemotherapy contraindications; Neutrophil absolute value ≥1.0×10^9 /L, PLT≥75×10^9 /L, hemoglobin ≥80g/L (except patients with lymphoma bone marrow infiltration);
5. At least one measurable lesion. For intrnodal lesions, they were defined as long diameter ≥1.5cm and short diameter ≥1.0cm; For r extranodal lesions, the length should be ≥1.0cm;

7. Liver function: TBIL≤1.5×ULN; ALT or AST ≤2.5 x ULN; Alkaline phosphatase ≤3×ULN in patients with non-bone invasion;

8. Kidney function: serum creatinine ≤1.5×ULN;

9. Excluding other major diseases, the heart function is normal;

10 Women and men of childbearing age and their spouses are willing to use adequate contraception throughout the study period, and women of childbearing age must have a negative serum pregnancy test within 7 days before the first dose;

11 Subjects voluntarily participated in the clinical trial, signed the informed consent form, and cooperated with the follow-up;

12. There is no other relevant treatment including traditional Chinese medicine (anti-tumor), immunotherapy, biologic therapy (except anti-bone metastasis and other symptoms);

Exclusion Criteria:

1. Patients with definite neuropathy or psychosis, including dementia or seizures, a history of psychotropic substance abuse and inability to abstinence, or other substantial lesions that may increase CNS toxicity;
2. Participating in other clinical trials or participating in other clinical investigators 4 weeks before enrollment (except those not receiving treatment);
3. Systemic autoimmune disease or immune deficiency;
4. Refusing to collect blood samples;
5. Allergic to any drug in the protocol;
6. Pregnant and lactating women;
7. Major diseases that can cause test interference and uncontrolled active infected persons;
8. Primary or secondary central tumor;
9. Contraindications to chemotherapy;
10. Not considered suitable for inclusion.
11. Known active bacterial, viral, fungal, mycobacterial, parasitic, or other infections (other than nail bed skin fungal infections) or any major systemic infection event requiring intravenous antibiotic treatment or hospitalization (other than neoplastic fever) within 4 weeks prior to enrollment;

13. Application of other antitumor therapies (such as radiotherapy, chemotherapy, hormone therapy, biotherapy, immunotherapy);

14. Other serious medical conditions that may limit the subject's participation in the study, such as uncontrolled diabetes; Severe cardiac insufficiency (NYHA grade II or above); Acute coronary syndrome in the last 6 months; Coronary revascularization such as stenting, cabG, and other cardiac and macrovascular procedures within the last 6 months; Severe arrhythmias include frequent ventricular premature, ventricular tachycardia, rapid atrial fibrillation/flutter, and severe bradycardia. Uncontrolled hypertension: systolic blood pressure >150mmHg, diastolic blood pressure >100mmHg. Gastric ulcers (those identified by the investigators as being at risk for perforation); Active autoimmune diseases (e.g. systemic lupus erythematosus, rheumatoid arthritis, multiple sclerosis, Sjogren's syndrome, autoimmune thrombocytopenia, etc.); Severe respiratory diseases (e.g. obstructive pulmonary disease and history of bronchospasm), etc.;

15. Hemophagocytic cell syndrome;

16. Hepatitis B surface antigen (HBsAg) or hepatitis B core antibody (HBcAb) was positive, and the peripheral blood hepatitis B virus (HBV) DNA titer was not within the normal reference range; Hepatitis C virus (HCV) antibody positive and HCV RNA positive in peripheral blood; Human immunodeficiency virus (HIV) antibody positive; Cytomegalovirus (CMV) DNA test positive; Who tested positive for syphilis.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A newly diagnosed patient with mantle cell lymphoma
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2022-08-12 (Actual); Primary Completion 2024-06-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
progression free survival（PFS） | two years
  progression free survival

SECONDARY OUTCOMES:
ORR | two years
  objective remission rate
CRR | two years
  complete remission rate
OS | two years
  overall survival
ADR | two years
  adverse drug reaction

CONTACTS AND LOCATIONS:
Overall Officials: Zhang Mingzhi Zhang, Principal Investigator — The First Affiliated Hospital of Zhengzhou University
Locations (1):
- Department of Oncology, The First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan, China